CLINICAL TRIAL: NCT04680351
Title: Evaluation of the Hemodynamic Effects of Transvenous Phrenic Stimulation
Acronym: HEMOSTIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 49RC20_0270
Record Dates: First submitted 2020-12-08; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Mechanical Ventilation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- phrenic stimulation (Experimental)
  Interventions: Procedure: phrenic stimulation

INTERVENTIONS:
Procedure: phrenic stimulation — measurements of the hemodynamic effects of phrenic stimulation

SUMMARY:
Mechanical ventilation is a cornerstone in the management of severe forms of pneumonia, acute respiratory distress syndrome. It provides essential oxygen to patients, ventilates the lungs but also has deleterious effects like any treatment, in particular by reducing cardiac output by reducing venous return. Mechanical ventilation also has effects on the diaphragm: diaphragmatic dysfunction. It is explained by a prolonged inactivity of this muscle with a reduction of muscle fibers that can settle down quickly, after only a few days of mechanical ventilation. This dysfunction results in a reduction in the latter's ability to generate intrathoracic pressure necessary for ventilation, slows the withdrawal of mechanical ventilation and lengthens the duration of stay in intensive care unit. To reduce this dysfunction, phrenic stimulation has been proposed as an alternative to remuscler the diaphragm thanks to electrodes located on a central venous catheter, also used to deliver the usual therapies in intensive care unit.

The HEMOSTIM study is interested in the effects of phrenic stimulation on regional ventilation, cardiac output and cerebral perfusion: investigator hypothesize that diaphragmatic stimulation allows an improvement of these parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patient included in RESCUE 3 study, interventional arm with phrenic stimulation
* Patient or family consent

Exclusion Criteria:

* Patient not affiliated or not benefiting from a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
measurement of integral time speed by cardiac transthoracic ultrasound | 1 minute
  to assess the effects of phrenic stimulation on cardiac output
Measurement of increased venous return gradient in percentage (variation between the value before phrenic stimulation and the value after phrenic stimulation) | 1 minute
  To specify the mechanisms of the effect of phrenic stimulation on cardiac output

SECONDARY OUTCOMES:
variation in ventilation distribution before and after phrenic stimulation measured in electrical impedance tomography | 1 minute
  To assess the effects of diaphragmatic stimulation on ventilation and pulmonary recruitment measured in electrical impedance tomography
Measurement of diaphragmatic stimulation on cerebral oxygenation evaluated by the Near infrared spectrometry technique | 1 minute

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Angers, Angers
  - APHP La Pitié-Salpêtrière, Paris

IPD SHARING:
Plan to Share IPD: No